CLINICAL TRIAL: NCT00709774
Title: Right Ventricular Septal Pacing for the Prevention of Left Ventricular Dysfunction in Patients With Atrio-Ventricular Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Osaka General Medical Center (Other)
Responsible Party: Yoshio Furukawa, Osaka General Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPaS-SvA
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-06

CONDITIONS: Atrio-Ventricular Block

INTERVENTIONS:
Device: Pacemaker Implantation — Implantation of right ventricular lead at septal or apex.

SUMMARY:
The aim of this study is to investigate the effects of the right ventricular septal pacing on left ventricular function compared with right ventricular apical pacing.

ELIGIBILITY:
Inclusion Criteria:

* the patients who need pacemaker implantation for atrio-ventricular block

Exclusion Criteria:

* Pregnancy, left ventricular dysfunction at the time of implantation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for the heart failure | 6 months

SECONDARY OUTCOMES:
incidence of atrial fibrillation | 6 months